CLINICAL TRIAL: NCT04132648
Title: Vasoconstrictor Responsiveness in Contracting Muscle of CKD: Influence of Acute Curcumin Supplementation
Brief Title: Curcumin and Exercise in Chronic Kidney Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left the Institution
Sponsor: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201907819
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Chronic Kidney Diseases; Blood Pressure; Hyperemia; Vasoconstriction
Keywords: CKD; Exercise; Vasoconstrictor Responsiveness
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperemia; Motor Activity | interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: Randomized Double-Blind Placebo-Controlled Crossover Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patient, providers, and the investigative team will all be blinded to the randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Curcumin (Experimental): Patients will receive curcumin (Longvida) 2000 mg one time prior to exercise trials
  Interventions: Drug: Curcumin
- Placebo (Placebo Comparator): Patients will receive placebo pill identical in appearance and taste to the supplement
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Curcumin — Oral supplement one time at 2,000 mg
  Other Names: Longvida
  Arms: Curcumin
Other: Placebo — Oral supplement one time at 2,000 mg
  Arms: Placebo

SUMMARY:
Chronic kidney disease (CKD) is associated with a pro-oxidative and pro-inflammatory state, and this is thought to contribute to a decrease in vascular function leading to greater cardiovascular disease (CVD) risk. Curcumin supplementation has been shown to reduce oxidative stress and improve endothelial function at rest in healthy older humans, although the magnitude of this effect remains unknown during exercise in CKD. The primary aim of this proposal is to determine whether exercising blood flow and vasoconstrictor responsiveness are improved as a result of acute oral supplementation with curcumin in patients with CKD. We hypothesize that: 1) acute curcumin supplementation will increase steady state exercise blood flow, and 2) reduce vasoconstriction induced by an acute sympathetic stimulus (cold pressor test) CKD.

DETAILED DESCRIPTION:
Active muscles require an optimal amount of local blood flow to meet the functional and metabolic demand of the exercising muscle. It is well known that maximal aerobic work capacity and exercise tolerance are reduced in CKD, contributing to functional impairment and loss of independence. A multitude of factors may be responsible for this outcome including reduced blood flow to active muscle beds brought on by greater levels of oxidative stress in CKD. Aging and some individuals with disease (coronary artery disease, hypertension, diabetes) exhibit elevated resting sympathetic nerve activity (SNA), leading to greater vasoconstriction and pressor responses during exercise. However, the magnitude of this effect remains unknown in CKD. Importantly, there are a lack of interventions aimed at improving blood flow and reduce sympathetic mediated vasoconstriction in patients with CKD.

Recent evidence in aging humans suggest that curcumin supplementation improves vascular function by reducing oxidative stress. However, it remains unknown whether acute curcumin supplementation can be regarded as an effective therapeutic strategy aimed at modulating exercise vasodilation and sympathetic mediated vasoconstriction in CKD. Understanding the mechanisms that impair vascular function within exercising muscle is important when understanding implications for systemic blood pressure regulation, cardiovascular disease and functional work capacity in CKD. Therefore, identifying a low cost, non-pharmaceutical intervention and its potential impact on improving vascular function in CKD is a priority in preventative cardiovascular disease medicine.

The present proposal aims to examine the effect of sympathetic vasoconstriction on the differential changes in exercising blood flow in response to acute oral supplementation with curcumin in patients with CKD.

ELIGIBILITY:
Inclusion Criteria for CKD subjects:

Age 45-80 years old CKD stage III and IV (estimated glomerular filtration rate: 15-60 mL/min/1.73m2) BMI <40 kg/m2-1 Able to give informed consent

Exclusion Criteria for CKD subjects will include answering yes to the following questions:

* Active participation in another study?
* Dialysis?
* End stage renal disease or kidney failure?
* Kidney transplant?
* Sever liver disease or transplant?
* Diabetes?
* Angina (i.e., chest discomfort/pain/pressure upon exertion)
* Severe congestive heart failure?
* Pacemaker/defibrillator?
* Heart arrhythmia (i.e. Atrial fibrillation/flutter)?
* Pregnant, breastfeeding, or unwilling to use adequate birth control?
* Active infection or antibiotic therapy?
* Immunosuppressive therapy within the last 3 months?
* History of stroke?
* Have you had a heart attack in the last 3 months?
* Have you taken curcumin in last 3 months?
* Current use of Hormone Replacement Therapy (if female)?
* Current smoker?
* Anemic (Hemoglobin count <9)?

Inclusion Criteria for healthy middle-age and older subjects:

Age 45-80 years old BMI <40 kg/m2 1 Able to give informed consent

Exclusion Criteria for health older subjects will include answering yes to the following questions:

* Chronic kidney disease?
* Hypertension?
* Asthma?
* Heart disease?
* Clinical depression?
* Autonomic disorders?
* Sleep apnea?
* Sever liver disease or transplant?
* Diabetes?
* Heart attack?
* Angina (i.e., chest discomfort/pain/pressure upon exertion)
* Severe systolic or congestive heart failure?
* Heart angioplasty/stent or bypass surgery?
* Heart valve surgery/replacement or valve disease?
* Pacemaker/defibrillator?
* Heart arrhythmia (i.e. Atrial fibrillation/flutter)?
* Pregnant, breastfeeding, or unwilling to use adequate birth control?
* Active infection or antibiotic therapy?
* Immunosuppressive therapy within the last 3 months?
* Have you taken curcumin in last 3 months?
* Current use of Hormone Replacement Therapy (if female)?
* Current smoker?
* Anemic (Hemoglobin count <9)?

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-15 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
%change forearm vascular condutance (FVC) | 2 hours
  Percentage reduction in FVC in response to acute sympathetic stimulus (cold pressor test; CPT)

SECONDARY OUTCOMES:
forearm blood flow (FBF) | 2 hours
  steady state FBF during forearm hand-grip exercise and CPT

IPD SHARING:
Plan to Share IPD: Undecided